CLINICAL TRIAL: NCT04404244
Title: Extraordinary Measures for Egyptian Children With Hemato-Oncological Disorders During COVID-19 Pandemic
Acronym: PedCan-COVID
Status: Completed | Type: Observational
Sponsor: Fatma Soliman Elsayed Ebeid, MD (Other)
Responsible Party: Sponsor-Investigator, Fatma Soliman Elsayed Ebeid, MD, Executive Director of Faculty of Medicine Ain Shams University Research Institute - Clinical Research Center, Ain Shams University
Organization: Ain Shams University (Other)
Other Study IDs: FMASU P25a/ 2020
Record Dates: First submitted 2020-05-25; First posted 2020-05-27 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Coronavirus COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective follow-up non-intervention study that will be carried out at Hematology/ Oncology Department, Children's hospital, Ain-Shams University, Cairo, Egypt. All followed-up children below 18 years with cancer during the one year study period from May 2020 till Apr 2021 either at the out-patients clinic or inpatient department will be recruited.

DETAILED DESCRIPTION:
Study Procedures:

On admission or during the outpatient visit:

1. Obtaining an informed consent .
2. Full medical history, concurrent medications, demographic data and epidemiological data (history of contact to a COVID-19 case, history of travel), will be obtained.
3. A thorough physical examination will be performed.
4. Body weight, height, BMI, vital signs (blood pressure, heart rate and temperature) and blood oxygen saturation) will be recorded.
5. Laboratory to perform the following tests:

Complete blood count with differential counts, COVID -19 reverse Transcription Polymerase Chain Reaction (RT-PCR) test by nasopharyngeal swab.

During admission:

Whenever unexplained fever and or respiratory symptoms developed or whenever COVID19 suspected to have the following to be performed:

1. Symptom developed that necessitates to repeat oropharyngeal and nasopharyngeal swab if indicated will be collected
2. Chest X-ray or CT chest will be recorded.
3. Laboratory to perform the following tests:

Complete blood count with differential counts,

COVID-19 RT-PCR test by oropharyngeal and nasopharyngeal swab:

C-reactive protein and serum ferritin level. Coagulation test; D. dimer, prothrombin time and INR. Routine bacteriological study, blood culture and other symptoms/signs based cultures will be recorded

On discharge:

* Date of discharge
* Period of admission
* Period of fever
* A thorough physical examination will be performed
* Record the outcome

ELIGIBILITY:
Inclusion Criteria:

1. Children below 18 years with malignancy either hematological or solid tumors or
2. Children below 18 years with hematological condition

Exclusion Criteria:

1. Patients or care-givers refusal to be enrolled in the study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All followed-up children below 18 years with with malignancy either hematological or solid tumors or hematological condition during the one year study period from May 2020 till Apr 2021 either at the out-patients clinic or inpatient department will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Incidence of COVID-19 among children with cancer | 12 months
  Measure the incidence of COVID-19 infection among children with cancer

SECONDARY OUTCOMES:
Families training | 12 months
  Families training about adhering to standard precautions for basic and respiratory hygiene to reduce the risk of transmission

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Ebeid, Principal Investigator — Excuitive Director of MARSI-CRC
Locations (1):
- Faculty of Medicine Ain Shams University Research Institute- Clinical Research Center, Cairo, Non-US, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ebeid FSE, Ragab IA, Elsherif NHK, Makkeyah S, Mostafa S, Eltonbary K, Matbouly S, Mostafa A, Goma H, Agwa SH, Hafez HM, Girgis S, El Gendy YG, El-Sayed MH. COVID-19 in Children With Cancer: A Single Low-Middle Income Center Experience. J Pediatr Hematol Oncol. 2021 Nov 1;43(8):e1077-e1081. doi: 10.1097/MPH.0000000000002025. PMID 33290293